CLINICAL TRIAL: NCT05275998
Title: A Phase 1b/2 Dose Escalation Study of the Safety, Pharmacokinetics, and Efficacy of the Combination of TMB-365 and TMB-380 in HIV-1 Infected Individuals Suppressed With Combination Antiretroviral Therapy
Brief Title: TMB-365 and TMB-380 in Suppressed HIV-1 Infected Individuals
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TMB-a21
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Results first posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection
Keywords: HIV-1 treatment, monoclonal antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sentinel Group 1 (Experimental): 10 HIV-1 infected subjects will receive one infusion of 2400 mg of each antibody, TMB-365 and TMB-380 and be followed for safety and pharmacokinetics. Oral suppressive cART will be continued throughout the course of the study participation.
  Interventions: Drug: TMB-365/TMB-380
- Sentinel Group 2 (Experimental): 10 HIV-1 infected subjects will receive one infusion of 3200 mg of each antibody, TMB-365 and TMB-380 and be followed for safety and pharmacokinetics. Oral suppressive cART will be continued throughout the course of the study participation.
  Interventions: Drug: TMB-365/TMB-380
- Sentinel Group 3 (Experimental): 10 HIV-1 infected subjects will receive one infusion of 4800 mg of each antibody, TMB-365 and TMB-380 and be followed for safety and pharmacokinetics. Oral suppressive cART will be continued throughout the course of the study participation.
  Interventions: Drug: TMB-365/TMB-380
- Core Group 1 (Experimental): 20 HIV-1 infected subjects will receive 4800 mg infusions of each antibody, TMB-365 and TMB-380 every 8 weeks and be followed for safety, pharmacokinetics, and ability to maintain antiviral activity. Oral suppressive cART will be discontinued for 24 weeks then resumed at week 24 with follow-up at week 28.
  Interventions: Drug: TMB-365/TMB-380

INTERVENTIONS:
Drug: TMB-365/TMB-380 — Monoclonal antibodies to be given intravenously
  Other Names: TMB-380 is also known as VRC07-523-LS

SUMMARY:
TMB-365 is a monoclonal antibody that binds to the CD4 receptor. TMB-380, aka VRC-07-523LS is a monoclonal antibody that binds to HIV. Both interfere with HIV entry. This study is designed to test various doses of the combination of the antibodies for safety and pharmacokinetics in suppressed subjects on cART. Once dosing is established based on safety and PK, the optimally dosed combinations will be assessed as maintenance therapy in HIV infected suppressed individuals discontinuing oral cART for 24 weeks.

DETAILED DESCRIPTION:
This study is a phase 1b / 2 adaptive open-label dose escalation study of the combination of TMB-365 and TMB-380. This adaptive study design will be comprised of Sentinel Groups (N=10) and Core Groups (N=20). Safety and pharmacokinetic (PK) data obtained from Sentinel group participants will guide the conduct of Core Group execution.

Participants will be HIV-infected and suppressed for at least 6 months on continuous daily oral combination antiretroviral therapy (cART). Continuous is defined as no more than 3 consecutive days of missed cART. There are three doses of each antibody being explored, 2400 mg, 3200 mg, and 4800 mg.

Sentinel Groups Sentinel Groups will be comprised of 10 cART suppressed HIV-1 infected volunteers who receive a single IV dose of the combination of TMB-365 and TMB-380 while continuing cART.

Sentinel Group 1 will be dosed with 2400 mg of each antibody and will continue daily oral cART throughout the screening, infusion, and post-infusion observation period of 12 and be assessed for safety and pharmacokinetics.

Sentinel group 2 will dose both antibodies at 3200 mg. The third sentinel group will dose both antibodies at 4800 mg.

Criteria for safety of a dose of either TMB-365 or TMB-380 include:

i) No SAEs probably or definitely due to TMB-365 or TMB-380 ii) No more than one Grade 3 or Grade 4 adverse event probably or definitely related to TMB-365 or TMB-380 at any dose level.

Toxicity evaluations will be guided by the DAIDS Table for Grading Severity of Adult and Pediatric Adverse Events Version 2.1. The Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0 scale will be used for assessment of any infusion reactions, or anaphylactic events.

PK targets:

i. TMB-365: serum levels >0.3 μg/mL ii. TMB-380: serum levels >65 μg/mL Should a dose of either antibody prove safe and at least 80% of subjects studied in a given Sentinel dose group meet specified safety and PK criteria, then a Core group of 20 subjects will be enrolled and treated with that dose of TMB-365 and TMB-380 as a stand-alone complete maintenance regimen for 24 weeks.

Safety must be established prior to any request for dose escalation to the next higher Sentinel dose group. A review of 14-day safety data in 7 of 10 subjects after infusion must be available for review prior to any request for dose escalation. Dose escalation may only occur with the approval of an independent Data Monitoring Committee (DMC).

The maximum dose of TMB-365 and TMB-380 that will be tested in Sentinel groups is 4800 mg.

The first 3 subjects in each Sentinel group will be treated at designated sites selected for demonstration of expertise in the use of monoclonal antibody therapy. Subjects will remain at the study site for 3 hours post-infusion for monitoring of vital signs every 15 minutes beginning 15 minutes prior to the infusion of TMB-365 and TMB-380 as well as observation for the presence of infusion reactions. Should the infusions be well tolerated and no Grade 3 or 4 AEs, or SAE's occur due to study drugs within 7 days of infusion, then the remaining 7 subjects in that group may be recruited/treated. These subjects will remain at study sites for 1 hour post-infusion for monitoring of vital signs and the presence of infusion reactions.

Core Group Subjects There will be one Core Group comprised of 40 cART suppressed HIV-1 infected volunteers and will receive multiple IV doses of the combination of TMB-365 and TMB-380 as a stand-alone maintenance regimen for 24 weeks. Oral cART will be restarted in the clinic at the Week 24 visit.

Core group participants will complete the study at Day 196, 4 weeks after reinstituting oral cART. Sentinel group participants at the same dosing level may be enrolled in a Core group if infusions are well tolerated and the subject is willing to discontinue oral cART.

Core Group study group 1 will begin with the doses of each antibody that prove safe and meet PK targets.

Regimen in Core Group participants based on PK modeling include:

TMB-365: 4800 mg q 8 weeks. TMB-380: 4800 mg q 8weeks. Sentinel Group participants that wish to participate in Core Groups must repeat all screening procedures including signing a second Informed Consent Form.

ELIGIBILITY:
Inclusion Criteria:Participants must meet all of the following criteria to be included in the study:

1. Male or female at least 18 years of age and no greater than 60 years on the day of Screening.
2. Asymptomatic HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by Geenius™ or a second antibody test by a method other than the initial rapid HIV and/or E/CIA test, or by HIV-1 antigen, plasma HIV-1 RNA viral load at or piror to screening.
3. On continuous suppressive cART for 6 months prior to screening with one documented HIV-1 RNA level below the level of detection within 3 months of screening. Continuous cART is defined as no interruptions greater than 3 consecutive days. cART is defined as a DHHS recommended regimen. Study participants should be on a stable regimen, at least 3 months.
4. Screening plasma HIV-1 RNA below the limit of detection.
5. CD4+ T cell count >350 cells/mm3
6. Laboratory values obtained within 30 days prior to the first dose:

   * Hemoglobin > 10.0 g/dL;
   * Platelet count ≥ 100,000/mm3;
   * Absolute neutrophil count ≥ 1,000/mm3;
   * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x upper limit of normal (ULN); and
   * Creatinine clearance (CrCl) of ≥ 50 mL/min.
7. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
8. In the opinion of the principal investigator or designee, has understood the information provided; written informed consent needs to be given before any study-related procedures are performed.
9. Females of childbearing potential, sexually active with a male sex partner, must agree to use one effective method of contraception from the time of signing the consent to completion of the study, and agree to pregnancy testing as per the Schedule of Events and Procedures. Females of childbearing potential are female participants who are not surgically sterile (no history of bilateral tubal ligation, hysterectomy, or bilateral salpingo-oophorectomy), are not postmenopausal (at least one year without menses), and are not otherwise sterile by medical evaluation.

   -

Exclusion Criteria:

Participants having or meeting any of the following conditions or characteristics will be excluded from the study:

1. Suppressed subjects who have not been on a stable DHHS recommended cART regimen for at least 3 months.
2. Receipt of any monoclonal antibody for the treatment or prevention of HIV infection except for Sentinel subjects eligible for enrollment into Core groups.
3. Suppressed subjects receiving cabotegravir and rilpivirine intramuscularly as maintenance therapy for HIV-1 infection.
4. Pregnant, planning a pregnancy during the trial period, or lactating.
5. Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation, or known allergy to a MAb.
6. Major psychiatric illness including any history of schizophrenia or severe psychosis, uncontrolled bipolar disorder requiring acute therapy, or suicide attempt in the previous three years.
7. Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to the first dose.
8. Receipt of immunomodulatory agents (e.g., interleukins, interferons, cyclosporine, high dose systemic corticosteroids), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 180 days prior to the first dose.
9. Any chronic or acute medical condition, including chronic Hepatits B infection, chronic Hepatitis C infection with viremia, and drug use and alcohol abuse, which in the opinion of the investigator would interfere with evaluation of the study drug.
10. Lack of adequate venous access.
11. Individuals who have experienced virologic failure during treatment with two or more cART treatment regimens and those being treated with regimens containing either ibalizumab, enfuvirtide, maraviroc, and fostemsavir. Note that a change in treatment regimen for intolerance does not meet criteria for virologic failure.

    -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Lalezari, MD, Principal Investigator — Quest Clinical Research
Locations (6):
- United States (6):
  - Quest Clinical Research, San Francisco, California
  - CAN Community Health, Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - North Texas Infectious Disease Consultants, Dallas, Texas
  - Crofoot Research Center, Inc., Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Group 1: 21 HIV-1 infected subjects will receive 4800 mg infusions of each antibody, TMB-365 and TMB-380 every 8 weeks and be followed for safety, pharmacokinetics, and ability to maintain antiviral activity. Oral suppressive cART will be discontinued for 24 weeks then resumed at week 24 with follow-up at week 28.
  TMB-365/TMB-380: Monoclonal antibodies to be given intravenously
Period: Overall Study
Arm/Group | Sentinel Group 1 | Sentinel Group 2 | Sentinel Group 3 | Core Group 1
Started | 10 | 10 | 10 | 21
Completed | 10 | 10 | 9 | 18
Not Completed | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study subjects are all HIV-infected, cART treated and suppressed on therapy for at least 6 months
Groups:
- Total: Total of all reporting groups
Arm/Group | Sentinel Group 1 | Sentinel Group 2 | Sentinel Group 3 | Core Group 1 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 21 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (7.9) | 43.1 (12.1) | 44 (10.1) | 49.3 (12.4) | 46.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 3
  Male | 10 | 9 | 9 | 20 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 5 | 11
  White | 7 | 6 | 7 | 14 | 34
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of TMB-365 and TMB-380 Given Intravenously (Sentinel and Core)
Description: Grade 3, Grade 4, Serious Adverse reactions related to TMB-365 and TMB-380 infusions
Time Frame: 12 weeks (Sentinel Group 1), 16 weeks (Sentinel Group 2, 3), 28 weeks (Core Group)
Population: Target enrollment in Core Group 1 is 20 participants. 21 were enrolled as one subject developed a serious medical condition between screen and baseline and was replaced. Therefore Core Group 1 consists of 20 evaluable participants.
Measure: Count of Participants; unit: Participants
Groups:
- Core Group 1: 20 HIV-1 infected subjects will receive 4800 mg infusions of each antibody, TMB-365 and TMB-380 every 8 weeks and be followed for safety, pharmacokinetics, and ability to maintain antiviral activity. Oral suppressive cART will be discontinued for 24 weeks then resumed at week 24 with follow-up at week 52.
  TMB-365/TMB-380: Monoclonal antibodies to be given intravenously
Arm/Group | Sentinel Group 1 | Sentinel Group 2 | Sentinel Group 3 | Core Group 1
Number analyzed (Participants) | 10 | 10 | 10 | 20
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Pharmacokinetics of a Single Dose TMB-365 Given Intravenously (Sentinel)
Description: In the Sentinel Group, participants received a single dose of TMB-365 and TMB-380 at 2400 mg, 3200 mg, or 4800 mg each. TMB-365 concentrations were measured using a validated ELISA, and the Week 8 concentration was used to guide dose selection for the Core Group.
Time Frame: Week 8
Population: One participant enrolled in Sentinel Group 3 was erroneously dosed with 1600 mg and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sentinel Group 1 | Sentinel Group 2 | Sentinel Group 3
Number analyzed (Participants) | 10 | 10 | 9
mcg/mL | 0.50 (1.23) | 1.91 (3.19) | 15.13 (13.45)

3. Primary Outcome: Pharmacokinetics of TMB-365 Given Intravenously Every 8 Weeks (Core)
Description: Core Group participants received 4800 mg every 8 weeks.TMB-365 concentrations were measured using a validated ELISA. Trough concentrations are reported.
Time Frame: Week 8, 16, and 24
Population: The Core Group enrolled 21 participants (one discontinued and was replaced), and 20 were considered evaluable. Two discontinued immediately after the Week 8 infusion, and one had no Week 24 data.
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Core Group: 21 HIV-1 infected subjects will receive 4800 mg infusions of each antibody, TMB-365 and TMB-380 every 8 weeks and be followed for safety, pharmacokinetics, and ability to maintain antiviral activity. Oral suppressive cART will be discontinued for 24 weeks then resumed at week 24 with follow-up at week 28.
  TMB-365/TMB-380: Monoclonal antibodies to be given intravenously
Arm/Group | Core Group
Number analyzed (Participants) | 20
mcg/mL
  Week 8 pre-dose concentration | 29.54 (30.18)
  Week 16 pre-dose concentration: number analyzed (Participants) | 18
  Week 16 pre-dose concentration | 29.12 (31.25)
  Week 24 trough concentration: number analyzed (Participants) | 17
  Week 24 trough concentration | 29.11 (35.94)

4. Secondary Outcome: Resistance to TMB-365 and TMB-380 (Core)
Description: Phenotype and genotype of HIV-1 variants in study subjects who fail to maintain antiviral response on infusions of TMB-365 and TMB-380
Time Frame: 24 weeks
Population: Resistance testing was conducted only in Core participants with virologic failure. As no virologic failures were observed, no resistance analyses were performed. Sentinel Group participants received TMB-365 or TMB-380 while continuing cART; therefore, resistance was not assessed.
Measure: Count of Participants; unit: Participants
Groups:
- Core Group 1: 20 HIV-1 infected subjects will receive 4800 mg infusions of each antibody, TMB-365 and TMB-380 every 8 weeks for 24 weeks as maintenance therapy (oral cART discontinued). Individuals with virologic failure will be assessed by genotype and phenotype for resistance to TMB-365 and TMB-380
  TMB-365/TMB-380: Monoclonal antibodies to be given intravenously
Arm/Group | Core Group 1
Number analyzed (Participants) | 0
Participants | 0

5. Primary Outcome: Pharmacokinetics of a Single Dose TMB-380 Given Intravenously (Sentinel)
Description: In the Sentinel Group, participants received a single dose of TMB-365 and TMB-380 at 2400 mg, 3200 mg, or 4800 mg each. TMB-380 concentrations were measured using a validated ELISA, and the Week 8 concentration was used to guide dose selection for the Core Group.
Time Frame: Week 8
Population: One participant enrolled in Sentinel Group 3 was erroneously dosed with 1600 mg and was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Sentinel Group 1 | Sentinel Group 2 | Sentinel Group 3
Number analyzed (Participants) | 10 | 10 | 9
mcg/mL | 59.59 (14.59) | 63.05 (16.47) | 86.43 (24.09)

6. Primary Outcome: Pharmacokinetics of TMB-380 Given Intravenously Every 8 Weeks (Core)
Description: Core Group participants received 4800 mg every 8 weeks.TMB-380 concentrations were measured using a validated ELISA. Trough concentrations are reported.
Time Frame: Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Core Group 1
Number analyzed (Participants) | 20
mcg/mL
  Week 8 pre-dose concentration | 83.72 (25.13)
  Week 16 pre-dose concentration: number analyzed (Participants) | 18
  Week 16 pre-dose concentration | 91.48 (21.93)
  Week 24 trough concentration: number analyzed (Participants) | 17
  Week 24 trough concentration | 107.12 (28.44)

7. Primary Outcome: Antiviral Activity of the Combination of TMB-365 in Combination With TMB-380 as Maintenance Therapy (Core)
Description: Plasma HIV-1 level below 50 copies/mL in study subjects at week 24 during maintenance therapy with TMB-365/TMB-380 infusions in Core Subjects only.
Time Frame: Week 24
Population: The Core Group enrolled 21 participants (one discontinued and was replaced), and 20 were considered evaluable. Two discontinued prematurely and one had no Week 24 data. The Sentinel Group participants received TMB-365 and TMB-380 while continuing cART, so antiviral activity was not assessed.
Measure: Count of Participants; unit: Participants
Groups:
- Core Group 1: 20 HIV-1 infected subjects will receive 4800 mg infusions of each antibody, TMB-365 and TMB-380 every 8 weeks and monitored for continued suppression of viral replication. Oral suppressive cART will be discontinued for 24 weeks then resumed at week 24 with follow-up at week 28.
  TMB-365/TMB-380: Monoclonal antibodies to be given intravenously
Arm/Group | Core Group 1
Number analyzed (Participants) | 17
Participants | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study which included a screening period of 6 weeks, 12 weeks for the 2400 mg and 3200 mg single dose group, 16 weeks for the 4800 mg single dose group, and 28 weeks for the 4800 mg multiple dose group (infusions for 24 weeks and 4 weeks of follow up)
Description: Adverse event reporting definitions do not differ from that described by clinicaltrials.gov
Arm/Group | Sentinel Group 1 | Sentinel Group 2 | Sentinel Group 3 | Core Group 1
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/21
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10 | 5/10 | 14/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Group 1 (N=10) | Sentinel Group 2 (N=10) | Sentinel Group 3 (N=10) | Core Group 1 (N=21)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4)
papules (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
attention deficit disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
syphilis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
streptococcal pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
oral pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Multi-Center Study Data are sponsor's property and sponsor must authorize publication. Sponsor and PIs together determine how a manuscript is written, edited and the publication to which it is submitted. Sponsor has final determination in these matters. PIs may publish or discuss their own study data with sponsor review at least 30 days in advance. Sponsor may require deletion of sponsor's confidential information and correction of inaccuracies, and request an embargo up to 60 additional days.

DOCUMENTS (2):
  • Study Protocol (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT05275998/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT05275998/SAP_001.pdf